CLINICAL TRIAL: NCT00004732
Title: Carotid Revascularization Endarterectomy Versus Stenting Trial (CREST)
Brief Title: Carotid Revascularization Endarterectomy Versus Stenting Trial
Acronym: CREST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0119970017; R01NS038384 (NIH)
Record Dates: First submitted 2000-02-25; First posted 2000-02-28 (Estimated); Results first posted 2013-12-10 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Atherosclerosis; Stroke; Carotid Stenosis; Cerebral Infarction; Myocardial Infarction
Keywords: angioplasty; asymptomatic; atherosclerosis; carotid endarterectomy; carotid stenting; CREST; Cerebral Infarction; device; intervention; restenosis; revascularization; stenosis; stent; stroke; symptomatic; surgery; transient ischemic attack
MeSH Terms: conditions — Atherosclerosis; Stroke; Carotid Stenosis; Cerebral Infarction; Myocardial Infarction; Constriction, Pathologic; Ischemic Attack, Transient | interventions — Endarterectomy, Carotid

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Carotid Artery Endarterectomy (CEA) (Active Comparator): Carotid endarterectomy is surgery to remove plaque buildup that causes narrowing (stenosis) in the carotid artery.
  Interventions: Procedure: Carotid Endarterectomy (CEA)
- Carotid Artery Stenting (CAS) (Active Comparator): Carotid artery stenting (CAS) is a procedure used to open narrowed carotid arteries. During the procedure, a small, expandable wire tube called a stent is permanently inserted into the carotid artery.
  Interventions: Device: Carotid Artery Stenting (CAS)

INTERVENTIONS:
Procedure: Carotid Endarterectomy (CEA) — CEA involves a neck incision and physical removal of the plaque from the inside of the carotid artery.
  Arms: Carotid Artery Endarterectomy (CEA)
Device: Carotid Artery Stenting (CAS) — CAS involves insertion of a catheter or tube into an artery in the groin and then threading the catheter through the arteries of the body to the location of the plaque within the carotid artery in the neck. A stent is then placed to cover the plaque and hold the artery open. Participants randomized to this arm of the trial were treated using the RX Acculink Carotid Stent with or without the RX Accunet Embolic Protection Device.
  Other Names: Angioplasty of carotid artery and stent placement.
  Arms: Carotid Artery Stenting (CAS)

SUMMARY:
The purpose of the Carotid Revascularization Endarterectomy versus Stenting Trial (CREST) is to compare the relatively new procedure of stent-assisted carotid angioplasty (CAS) to the traditional and accepted surgical approach of carotid endarterectomy (CEA) for the treatment of carotid artery stenosis to prevent recurrent strokes in those patients who have had a TIA (transient ischemic attack) or a mild stroke within the past 6 months (symptomatic) and in those patients who have not had any symptoms within the past 6 months (asymptomatic).

DETAILED DESCRIPTION:
The primary aim of the Carotid Revascularization Endarterectomy versus Stenting Trial (CREST) is to contrast the relative effectiveness of carotid artery stenting (CAS) versus carotid endarterectomy (CEA) in preventing stroke, myocardial infarction, and death. Stents are medical devices approved and commonly used for treatment of heart disease. The stent that will be used in this trial is the Rapid Exchange(RX) ACCULINK(TM) Carotid Stent System, an elastic-like metal scaffold that is expanded inside a carotid artery to hold the vessel open.

The RX ACCUNET(TM) Embolic Protection System (an umbrella-like device that expands above the narrowed portion of the carotid artery) will be used in conjunction with the RX ACCULINK stent. The RX ACCUNET system is designed to capture embolic material that could break off from the narrowed area in the carotid artery while still allowing blood to flow through the vessel during the procedure. Embolic material could block blood flow to the arteries beyond the narrowing and be harmful to the brain. The RX ACCUNET System is closed and removed after the stent is placed.

CEA involves a neck incision and physical removal of the plaque from the inside of the artery. CAS involves insertion of a catheter or tube into an artery in the groin and then threading the catheter through the arteries of the body to the location of the plaque within the carotid artery in the neck. The stent is then placed to cover the plaque and hold the artery open. Participants will be randomly assigned to undergo either CAS or CEA, and all patients will receive best medical management, which includes treatment with aspirin, treatment of high blood pressure, and treatment of other stroke risk factors. Participants will be followed for up to ten years.

With the simplification of the protocol for long-term follow-up, the focus for secondary outcomes is to assess restenosis and viability of the procedure. Restenosis rates on an annual basis in both the endarterectomy and stenting arms of the study will be assessed using carotid duplex ultrasound exams performed annually (standard of care).

In addition to restenosis, the "viability" of the procedures will be assessed by the need (or lack of need) for repeat revascularization (either open surgical or endovascular) after the index procedure. The question "has a new carotid intervention been performed since last follow-up" will be asked at every contact with the patient. If answered positively, additional data will be collected on the appropriate case report forms(CRFs).

LINKAGE OF CREST COHORT WITH CENTERS FOR MEDICAID AND MEDICARE SERVICES(CMS) ADMINISTRATIVE DATA

The purpose of linking Medicare-eligible CREST participants with CMS data files is to assess patient outcomes and utilization of health care services. This plan to link in- and out-patient episodes of care using national Medicare data establishes a new resource that will enhance current follow-up strategies, as well as explore alternative strategies to ascertain patient outcomes for future clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic patients with recent neurological events (TIA or non-disabling stroke) with an associated carotid stenosis greater than or equal to 50% by angiography or greater than or equal to 70% by ultrasound or greater than or equal to 70% by Computed Tomography Angiography (CTA) or Magnetic Resonance Angiography (MRA) are eligible for randomization.
* Asymptomatic patients with no recent (in the last 6 months) neurological events referable to the study with artery and carotid stenosis (patients with symptoms beyond 180 days are considered asymptomatic) greater than or equal to 60% by angiography or greater than or equal to 70% by ultrasound or greater than or equal to 80% by CTA or MRA are eligible for randomization.

Exclusion Criteria:

* Conditions that: (1) interfere with the evaluation of endpoints, (2) are known to interfere with the completion of CEA or CAS, or (3) affect the likelihood of survival for the study period (4 years). Chronic atrial fibrillation and/or anti-coagulation or episodic atrial fibrillation within the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2502 (Actual)
Dates: Start 2000-12; Primary Completion 2011-02 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G. Brott, M.D., Principal Investigator — Mayo Clinic and Rutgers University
Locations (115):
- United States (106):
  - The Board of Trustees of the University of Alabama for the University of Alabama at Birmingham, Birmingham, Alabama
  - Dignity Health dba St. Joseph's Hospital & Medical Center, Phoenix, Arizona
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - The Arizona Board of Regents for the University of Arizona, Tucson, Arizona
  - Board of Trustees of the University of Arkansas, Little Rock, Arkansas
  - USC University Hospital & LA County Hospital, Los Angeles, California
  - The Regents of the University of California, Los Angeles, California
  - Kaiser Permanente Medical Center, San Diego, California
  - Northern California Institute for Research and Education, San Francisco, California
  - Catholic Healthcare West, Stockton, California
  - Christiana Care Health Services, Inc., Newark, Delaware
  - Morton Plant Hospital, Clearwater, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Leesburg Medical Center, Leesburg, Florida
  - Miami Cardiac & Vascular Institute of Baptist Hospital of Miami, Inc., Miami, Florida
  - Florida Hospital Neuroscience Institute, a division of Adventist Health System/Sunbelt, Inc., Orlando, Florida
  - Orlando Regional Medical Center, Orlando, Florida
  - University of South Florida Board of Trustees, Tampa, Florida
  - Piedmont Hospital/Fuqua Heart Center, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - St. Joseph's of Atlanta, Atlanta, Georgia
  - St. Joseph's Candler Health System, Savannah, Georgia
  - Norwestern Memorial Hospital, Chicago, Illinois
  - Alexian Brothers Specialty Group, Elk Grove Village, Illinois
  - Loyola University of Chicago, Maywood, Illinois
  - Peoria Radiology Research and Education, Peoria, Illinois
  - Prarie Cardiology-St. John's Hospital, Springfield, Illinois
  - Southern Illinois School of Medicine, Springfield, Illinois
  - Central Dupage Hospital, Winfield, Illinois
  - Lutheran Medical Group, LLC,, Fort Wayne, Indiana
  - Parkview Hospital, Inc., Fort Wayne, Indiana
  - St. Vincent's Hospital, Indianapolis, Indiana
  - Catholic Health Initiatives /Mercy Hospital Center, Des Moines, Iowa
  - Baptist Healthcare System, Inc., Lexington, Kentucky
  - Vascular Surgery Associates, Baton Rouge, Louisiana
  - Ochsner Foundation Hospital, New Orleans, Louisiana
  - Anne Arundel Health System Research Institute, Annapolis, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Adventist Healthcare, Inc., Takoma Park, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Steward St. Elizabeth's Medical Center of Boston, Inc., Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Womens Hospital, Inc., Boston, Massachusetts
  - Cape Cod Health Care, Inc.,, Hyannis, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - St. John Hospital and Medical Center, Detroit, Michigan
  - Michigan Vascular Research Center, Flint, Michigan
  - Spectrum Health Hospital, Grand Rapids, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Providence St. John Hopital, Southfield, Michigan
  - Michigan Heart & Vascular Institute/St. Joseph's Mercy Hospital, Ypsilanti, Michigan
  - North Memorial Health Care, Robbinsdale, Minnesota
  - Mayo Clinic Rochester/St. Mary's, Rochester, Minnesota
  - Mississippi Baptist Medical Center, Inc., Jackson, Mississippi
  - Heartland Physician Services, LLC, Kansas City, Missouri
  - Mercy Hospitals East Communities, St Louis, Missouri
  - St. Patrick's Hospital International Heart Institute of MT, Missoula, Montana
  - Dartmouth College and the constituent members of DARTMOUTH HITCHCOCK MEDICAL CENTER, Lebanon, New Hampshire
  - St. Michael's Medical Center, Newark, New Jersey
  - Center for Vascular Awareness, Inc., Albany, New York
  - Millard Fillmore SUNY Buffalo, Buffalo, New York
  - NYU School of Medicine, New York, New York
  - The Feinstein Institute for Medical Research, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Columbia Presbyterian, New York, New York
  - St. Francis Hospital, Port Washington, New York
  - University of Rochester, Rochester, New York
  - Richmond University Medical Center, Staten Island, New York
  - Westchester Medical Center, Valhalla, New York
  - UNC at Chapel Hill, Chapel Hill, North Carolina
  - The Charlotte-Mecklenburg Hospital Authority, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Forsyth Radiological Associates, Winston-Salem, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - The Cleveland Clinic Lerner College Of Medicine of CWRU, Cleveland, Ohio
  - Midwest Ohio Health Research Institute, Columbus, Ohio
  - The Toledo Hospital, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Oklahoma Foundation for Cardiovascular Research, Oklahoma City, Oklahoma
  - Rogue Valley Medical Center, Medford, Oregon
  - Oregon Health Science University, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Heritage Valley Medical Group, Beaver, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Allegheny Singer Research Institute, Pittsburgh, Pennsylvania
  - UPMC Presbyterian Shadyside, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - South Carolina Heart Center, Columbia, South Carolina
  - Metro Knoxville HMA, Knoxville, Tennessee
  - Baptist Memorial Hospital, Memphis, Tennessee
  - The University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - UT Houston Memorial, Houston, Texas
  - Scott & White Memorial Hospital, Temple, Texas
  - Intermountain Health Services, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Swedish Health Services, Seattle, Washington
  - Providence Health & Services - Washington, Spokane, Washington
  - Charleston Area Medical Center, Charleston, West Virginia
  - Marshfield Clinic, Marshfield, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin
- Canada (9):
  - Governors of the University of Calgary and the Calgary Health Region, Calgary, Alberta
  - The University of British Columbia and The Vancouver Coastal Health Authority, Vancouver, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - The Credit Valley Hospital and Trillium Health Centre, Mississauga, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Lawson Health Research Institute, Toronto, Ontario
  - CHU de Québec, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hopkins LN, Roubin GS, Chakhtoura EY, Gray WA, Ferguson RD, Katzen BT, Rosenfield K, Goldstein J, Cutlip DE, Morrish W, Lal BK, Sheffet AJ, Tom M, Hughes S, Voeks J, Kathir K, Meschia JF, Hobson RW 2nd, Brott TG. The Carotid Revascularization Endarterectomy versus Stenting Trial: credentialing of interventionalists and final results of lead-in phase. J Stroke Cerebrovasc Dis. 2010 Mar;19(2):153-62. doi: 10.1016/j.jstrokecerebrovasdis.2010.01.001. PMID 20189092
- [Background] Howard VJ, Voeks JH, Lutsep HL, Mackey A, Milot G, Sam AD 2nd, Tom M, Hughes SE, Sheffet AJ, Longbottom M, Avery JB, Hobson RW 2nd, Brott TG. Does sex matter? Thirty-day stroke and death rates after carotid artery stenting in women versus men: results from the Carotid Revascularization Endarterectomy versus Stenting Trial (CREST) lead-in phase. Stroke. 2009 Apr;40(4):1140-7. doi: 10.1161/STROKEAHA.108.541847. Epub 2009 Feb 10. PMID 19211486
- [Background] Sheffet AJ, Roubin G, Howard G, Howard V, Moore W, Meschia JF, Hobson RW 2nd, Brott TG. Design of the Carotid Revascularization Endarterectomy vs. Stenting Trial (CREST). Int J Stroke. 2010 Feb;5(1):40-6. doi: 10.1111/j.1747-4949.2009.00405.x. PMID 20088993
- [Background] Lal BK, Brott TG. The Carotid Revascularization Endarterectomy vs. Stenting Trial completes randomization: lessons learned and anticipated results. J Vasc Surg. 2009 Nov;50(5):1224-31. doi: 10.1016/j.jvs.2009.09.003. PMID 19878793
- [Background] Hobson RW 2nd, Brott TG, Roubin GS, Silver FL, Barnett HJ. Carotid artery stenting: meeting the recruitment challenge of a clinical trial. Stroke. 2005 Jun;36(6):1314-5. doi: 10.1161/01.STR.0000165919.26944.05. Epub 2005 Apr 28. No abstract available. PMID 15860747
- [Background] Hobson RW 2nd, Howard VJ, Roubin GS, Brott TG, Ferguson RD, Popma JJ, Graham DL, Howard G; CREST Investigators. Carotid artery stenting is associated with increased complications in octogenarians: 30-day stroke and death rates in the CREST lead-in phase. J Vasc Surg. 2004 Dec;40(6):1106-11. doi: 10.1016/j.jvs.2004.10.022. PMID 15622363
- [Background] Hobson RW 2nd, Howard VJ, Roubin GS, Ferguson RD, Brott TG, Howard G, Sheffet AJ, Roberts J, Hopkins LN, Moore WS; CREST. Credentialing of surgeons as interventionalists for carotid artery stenting: experience from the lead-in phase of CREST. J Vasc Surg. 2004 Nov;40(5):952-7. doi: 10.1016/j.jvs.2004.08.039. PMID 15557910
- [Background] Hobson RW 2nd, Howard VJ, Brott TG, Howard G, Roubin GS, Ferguson RD; For the CREST Executive Committee. Organizing the Carotid Revascularization Endarterectomy versus Stenting Trial (CREST): National Institutes of Health, Health Care Financing Administration, and industry funding. Curr Control Trials Cardiovasc Med. 2001 Jul 13;2(4):160-164. doi: 10.1186/cvm-2-4-160. PMID 11806790
- [Background] Hobson RW 2nd, Brott T, Ferguson R, Roubin G, Moore W, Kuntz R, Howard G, Ferguson J. CREST: carotid revascularization endarterectomy versus stent trial. Cardiovasc Surg. 1997 Oct;5(5):457-8. doi: 10.1016/s0967-2109(97)00048-3. No abstract available. PMID 9464598
- [Result] Brott TG, Hobson RW 2nd, Howard G, Roubin GS, Clark WM, Brooks W, Mackey A, Hill MD, Leimgruber PP, Sheffet AJ, Howard VJ, Moore WS, Voeks JH, Hopkins LN, Cutlip DE, Cohen DJ, Popma JJ, Ferguson RD, Cohen SN, Blackshear JL, Silver FL, Mohr JP, Lal BK, Meschia JF; CREST Investigators. Stenting versus endarterectomy for treatment of carotid-artery stenosis. N Engl J Med. 2010 Jul 1;363(1):11-23. doi: 10.1056/NEJMoa0912321. Epub 2010 May 26. PMID 20505173
- [Result] Mantese VA, Timaran CH, Chiu D, Begg RJ, Brott TG; CREST Investigators. The Carotid Revascularization Endarterectomy versus Stenting Trial (CREST): stenting versus carotid endarterectomy for carotid disease. Stroke. 2010 Oct;41(10 Suppl):S31-4. doi: 10.1161/STROKEAHA.110.595330. PMID 20876500
- [Result] Silver FL, Mackey A, Clark WM, Brooks W, Timaran CH, Chiu D, Goldstein LB, Meschia JF, Ferguson RD, Moore WS, Howard G, Brott TG; CREST Investigators. Safety of stenting and endarterectomy by symptomatic status in the Carotid Revascularization Endarterectomy Versus Stenting Trial (CREST). Stroke. 2011 Mar;42(3):675-80. doi: 10.1161/STROKEAHA.110.610212. Epub 2011 Feb 9. PMID 21307169
- [Result] Blackshear JL, Cutlip DE, Roubin GS, Hill MD, Leimgruber PP, Begg RJ, Cohen DJ, Eidt JF, Narins CR, Prineas RJ, Glasser SP, Voeks JH, Brott TG; CREST Investigators. Myocardial infarction after carotid stenting and endarterectomy: results from the carotid revascularization endarterectomy versus stenting trial. Circulation. 2011 Jun 7;123(22):2571-8. doi: 10.1161/CIRCULATIONAHA.110.008250. Epub 2011 May 23. PMID 21606394
- [Result] Vilain KR, Magnuson EA, Li H, Clark WM, Begg RJ, Sam AD 2nd, Sternbergh WC 3rd, Weaver FA, Gray WA, Voeks JH, Brott TG, Cohen DJ; CREST Investigators. Costs and cost-effectiveness of carotid stenting versus endarterectomy for patients at standard surgical risk: results from the Carotid Revascularization Endarterectomy Versus Stenting Trial (CREST). Stroke. 2012 Sep;43(9):2408-16. doi: 10.1161/STROKEAHA.112.661355. Epub 2012 Jul 19. PMID 22821614
- [Result] Lal BK, Beach KW, Roubin GS, Lutsep HL, Moore WS, Malas MB, Chiu D, Gonzales NR, Burke JL, Rinaldi M, Elmore JR, Weaver FA, Narins CR, Foster M, Hodgson KJ, Shepard AD, Meschia JF, Bergelin RO, Voeks JH, Howard G, Brott TG; CREST Investigators. Restenosis after carotid artery stenting and endarterectomy: a secondary analysis of CREST, a randomised controlled trial. Lancet Neurol. 2012 Sep;11(9):755-63. doi: 10.1016/S1474-4422(12)70159-X. Epub 2012 Aug 2. PMID 22857850
- [Result] Hill MD, Brooks W, Mackey A, Clark WM, Meschia JF, Morrish WF, Mohr JP, Rhodes JD, Popma JJ, Lal BK, Longbottom ME, Voeks JH, Howard G, Brott TG; CREST Investigators. Stroke after carotid stenting and endarterectomy in the Carotid Revascularization Endarterectomy versus Stenting Trial (CREST). Circulation. 2012 Dec 18;126(25):3054-61. doi: 10.1161/CIRCULATIONAHA.112.120030. Epub 2012 Nov 16. PMID 23159552
- [Result] Timaran CH, Mantese VA, Malas M, Brown OW, Lal BK, Moore WS, Voeks JH, Brott TG; CREST Investigators. Differential outcomes of carotid stenting and endarterectomy performed exclusively by vascular surgeons in the Carotid Revascularization Endarterectomy versus Stenting Trial (CREST). J Vasc Surg. 2013 Feb;57(2):303-8. doi: 10.1016/j.jvs.2012.09.014. Epub 2012 Dec 20. PMID 23265585
- [Derived] Matsumura JS, Hanlon BM, Rosenfield K, Voeks JH, Howard G, Roubin GS, Brott TG. Treatment of carotid stenosis in asymptomatic, nonoctogenarian, standard risk patients with stenting versus endarterectomy trials. J Vasc Surg. 2022 Apr;75(4):1276-1283.e1. doi: 10.1016/j.jvs.2021.10.020. Epub 2021 Oct 22. PMID 34695552
- [Derived] Howard VJ, Algra A, Howard G, Bonati LH, de Borst GJ, Bulbulia R, Calvet D, Eckstein HH, Fraedrich G, Greving JP, Halliday A, Hendrikse J, Jansen O, Brown MM, Mas JL, Ringleb PA, Brott TG; Carotid Stenosis Trialists' Collaboration. Absence of Consistent Sex Differences in Outcomes From Symptomatic Carotid Endarterectomy and Stenting Randomized Trials. Stroke. 2021 Jan;52(2):416-423. doi: 10.1161/STROKEAHA.120.030184. Epub 2021 Jan 25. PMID 33493046
- [Derived] Muller MD, von Felten S, Algra A, Becquemin JP, Bulbulia R, Calvet D, Eckstein HH, Fraedrich G, Halliday A, Hendrikse J, Howard G, Gregson J, Jansen O, Brown MM, Mas JL, Brott TG, Ringleb PA, Bonati LH. Secular Trends in Procedural Stroke or Death Risks of Stenting Versus Endarterectomy for Symptomatic Carotid Stenosis. Circ Cardiovasc Interv. 2019 Aug;12(8):e007870. doi: 10.1161/CIRCINTERVENTIONS.119.007870. Epub 2019 Aug 5. PMID 31378071
- [Derived] Moore WS, Voeks JH, Roubin GS, Clark WM, Howard VJ, Jones MR, Brott TG; CREST Investigators. Duration of asymptomatic status and outcomes following carotid endarterectomy and carotid artery stenting in the Carotid Revascularization Endarterectomy vs Stenting Trial. J Vasc Surg. 2019 Jun;69(6):1797-1800. doi: 10.1016/j.jvs.2018.09.054. Epub 2019 Jan 8. PMID 30630649
- [Derived] Jones MR, Howard G, Roubin GS, Blackshear JL, Cohen DJ, Cutlip DE, Leimgruber PP, Rhodes D, Prineas RJ, Glasser SP, Lal BK, Voeks JH, Brott TG; CREST Investigators. Periprocedural Stroke and Myocardial Infarction as Risks for Long-Term Mortality in CREST. Circ Cardiovasc Qual Outcomes. 2018 Nov;11(11):e004663. doi: 10.1161/CIRCOUTCOMES.117.004663. PMID 30571337
- [Derived] Lal BK, Roubin GS, Jones M, Clark W, Mackey A, Hill MD, Voeks JH, Howard G, Hobson RW 2nd, Brott TG. Influence of multiple stents on periprocedural stroke after carotid artery stenting in the Carotid Revascularization Endarterectomy versus Stent Trial (CREST). J Vasc Surg. 2019 Mar;69(3):800-806. doi: 10.1016/j.jvs.2018.06.221. Epub 2018 Dec 4. PMID 30527940
- [Derived] Muller MD, von Felten S, Algra A, Becquemin JP, Brown M, Bulbulia R, Calvet D, Eckstein HH, Fraedrich G, Halliday A, Hendrikse J, Gregson J, Howard G, Jansen O, Mas JL, Brott TG, Ringleb PA, Bonati LH; Carotid Stenosis Trialists' Collaboration. Immediate and Delayed Procedural Stroke or Death in Stenting Versus Endarterectomy for Symptomatic Carotid Stenosis. Stroke. 2018 Nov;49(11):2715-2722. doi: 10.1161/STROKEAHA.118.020684. PMID 30355202
- [Derived] Sheffet AJ, Howard G, Sam A, Jamil Z, Weaver F, Chiu D, Voeks JH, Howard VJ, Hughes SE, Flaxman L, Longbottom ME, Brott TG; CREST Investigators. Challenge and Yield of Enrolling Racially and Ethnically Diverse Patient Populations in Low Event Rate Clinical Trials. Stroke. 2018 Jan;49(1):84-89. doi: 10.1161/STROKEAHA.117.018063. Epub 2017 Nov 30. PMID 29191852
- [Derived] Rantner B, Kollerits B, Roubin GS, Ringleb PA, Jansen O, Howard G, Hendrikse J, Halliday A, Gregson J, Eckstein HH, Calvet D, Bulbulia R, Bonati LH, Becquemin JP, Algra A, Brown MM, Mas JL, Brott TG, Fraedrich G; Carotid Stenosis Trialists' Collaboration. Early Endarterectomy Carries a Lower Procedural Risk Than Early Stenting in Patients With Symptomatic Stenosis of the Internal Carotid Artery: Results From 4 Randomized Controlled Trials. Stroke. 2017 Jun;48(6):1580-1587. doi: 10.1161/STROKEAHA.116.016233. Epub 2017 Apr 28. PMID 28455318
- [Derived] Brott TG, Howard G, Roubin GS, Meschia JF, Mackey A, Brooks W, Moore WS, Hill MD, Mantese VA, Clark WM, Timaran CH, Heck D, Leimgruber PP, Sheffet AJ, Howard VJ, Chaturvedi S, Lal BK, Voeks JH, Hobson RW 2nd; CREST Investigators. Long-Term Results of Stenting versus Endarterectomy for Carotid-Artery Stenosis. N Engl J Med. 2016 Mar 17;374(11):1021-31. doi: 10.1056/NEJMoa1505215. Epub 2016 Feb 18. PMID 26890472
- [Derived] Moore WS, Popma JJ, Roubin GS, Voeks JH, Cutlip DE, Jones M, Howard G, Brott TG; CREST Investigators. Carotid angiographic characteristics in the CREST trial were major contributors to periprocedural stroke and death differences between carotid artery stenting and carotid endarterectomy. J Vasc Surg. 2016 Apr;63(4):851-7, 858.e1. doi: 10.1016/j.jvs.2015.08.119. Epub 2015 Nov 21. PMID 26610643
- [Derived] Meschia JF, Hopkins LN, Altafullah I, Wechsler LR, Stotts G, Gonzales NR, Voeks JH, Howard G, Brott TG. Time From Symptoms to Carotid Endarterectomy or Stenting and Perioperative Risk. Stroke. 2015 Dec;46(12):3540-2. doi: 10.1161/STROKEAHA.115.011123. Epub 2015 Oct 22. PMID 26493675
- [Derived] Voeks JH, Howard G, Roubin G, Farb R, Heck D, Logan W, Longbottom M, Sheffet A, Meschia JF, Brott TG. Mediators of the Age Effect in the Carotid Revascularization Endarterectomy Versus Stenting Trial (CREST). Stroke. 2015 Oct;46(10):2868-73. doi: 10.1161/STROKEAHA.115.009516. Epub 2015 Sep 8. PMID 26351359
- [Derived] Howard G, Hopkins LN, Moore WS, Katzen BT, Chakhtoura E, Morrish WF, Ferguson RD, Hye RJ, Shawl FA, Harrigan MR, Voeks JH, Howard VJ, Lal BK, Meschia JF, Brott TG. Temporal Changes in Periprocedural Events in the Carotid Revascularization Endarterectomy Versus Stenting Trial. Stroke. 2015 Aug;46(8):2183-9. doi: 10.1161/STROKEAHA.115.008898. Epub 2015 Jul 14. PMID 26173731
- [Derived] Sheffet AJ, Voeks JH, Mackey A, Brooks W, Clark WM, Hill MD, Howard VJ, Hughes SE, Tom M, Longbottom ME, Brott TG; CREST Investigators. Characteristics of participants consenting versus declining follow-up for up to 10 years in a randomized clinical trial. Clin Trials. 2015 Dec;12(6):657-63. doi: 10.1177/1740774515590807. Epub 2015 Jun 29. PMID 26122922
- [Derived] Malas M, Glebova NO, Hughes SE, Voeks JH, Qazi U, Moore WS, Lal BK, Howard G, Llinas R, Brott TG. Effect of patching on reducing restenosis in the carotid revascularization endarterectomy versus stenting trial. Stroke. 2015 Mar;46(3):757-61. doi: 10.1161/STROKEAHA.114.007634. Epub 2015 Jan 22. PMID 25613307
- [Derived] Meschia JF, Voeks JH, Leimgruber PP, Mantese VA, Timaran CH, Chiu D, Demaerschalk BM, Howard VJ, Hughes SE, Longbottom M, Howard AG, Brott TG. Management of vascular risk factors in the Carotid Revascularization Endarterectomy Versus Stenting Trial (CREST). J Am Heart Assoc. 2014 Nov 26;3(6):e001180. doi: 10.1161/JAHA.114.001180. PMID 25428209
- [Derived] Gonzales NR, Demaerschalk BM, Voeks JH, Tom M, Howard G, Sheffet AJ, Garcia L, Clair DG, Barr J, Orlow S, Brott TG; CREST Investigators. Complication rates and center enrollment volume in the carotid revascularization endarterectomy versus stenting trial. Stroke. 2014 Nov;45(11):3320-4. doi: 10.1161/STROKEAHA.114.006228. Epub 2014 Sep 25. PMID 25256180
- [Derived] Howard G, Voeks JH, Meschia JF, Howard VJ, Brott TG. Picking the good apples: statistics versus good judgment in choosing stent operators for a multicenter clinical trial. Stroke. 2014 Nov;45(11):3325-9. doi: 10.1161/STROKEAHA.114.006807. Epub 2014 Sep 11. PMID 25213339
- [Derived] Sheffet AJ, Flaxman L, Tom M, Hughes SE, Longbottom ME, Howard VJ, Marler JR, Brott TG; CREST Investigators. Financial management of a large multisite randomized clinical trial. Int J Stroke. 2014 Aug;9(6):811-3. doi: 10.1111/ijs.12259. Epub 2014 Mar 24. PMID 24661748
- [Derived] Zierler RE, Beach KW, Bergelin RO, Lal BK, Moore WS, Roubin GS, Voeks JH, Brott TG; CREST Investigators. Agreement between site-reported and ultrasound core laboratory results for duplex ultrasound velocity measurements in the Carotid Revascularization Endarterectomy versus Stenting Trial. J Vasc Surg. 2014 Jan;59(1):2-7. doi: 10.1016/j.jvs.2013.06.071. Epub 2013 Sep 19. PMID 24055515
- [Derived] Habersberger J, Brott TG, Roubin GS. Carotid artery stenting: a clinical update. Curr Opin Cardiol. 2012 Nov;27(6):565-71. doi: 10.1097/HCO.0b013e3283587506. PMID 22941123
- [Derived] Voeks JH, Howard G, Roubin GS, Malas MB, Cohen DJ, Sternbergh WC 3rd, Aronow HD, Eskandari MK, Sheffet AJ, Lal BK, Meschia JF, Brott TG; CREST Investigators. Age and outcomes after carotid stenting and endarterectomy: the carotid revascularization endarterectomy versus stenting trial. Stroke. 2011 Dec;42(12):3484-90. doi: 10.1161/STROKEAHA.111.624155. Epub 2011 Oct 6. PMID 21980205
- [Derived] Cohen DJ, Stolker JM, Wang K, Magnuson EA, Clark WM, Demaerschalk BM, Sam AD Jr, Elmore JR, Weaver FA, Aronow HD, Goldstein LB, Roubin GS, Howard G, Brott TG; CREST Investigators. Health-related quality of life after carotid stenting versus carotid endarterectomy: results from CREST (Carotid Revascularization Endarterectomy Versus Stenting Trial). J Am Coll Cardiol. 2011 Oct 4;58(15):1557-65. doi: 10.1016/j.jacc.2011.05.054. PMID 21958882
- [Derived] Chimowitz MI, Lynn MJ, Derdeyn CP, Turan TN, Fiorella D, Lane BF, Janis LS, Lutsep HL, Barnwell SL, Waters MF, Hoh BL, Hourihane JM, Levy EI, Alexandrov AV, Harrigan MR, Chiu D, Klucznik RP, Clark JM, McDougall CG, Johnson MD, Pride GL Jr, Torbey MT, Zaidat OO, Rumboldt Z, Cloft HJ; SAMMPRIS Trial Investigators. Stenting versus aggressive medical therapy for intracranial arterial stenosis. N Engl J Med. 2011 Sep 15;365(11):993-1003. doi: 10.1056/NEJMoa1105335. Epub 2011 Sep 7. PMID 21899409
- [Derived] Howard VJ, Lutsep HL, Mackey A, Demaerschalk BM, Sam AD 2nd, Gonzales NR, Sheffet AJ, Voeks JH, Meschia JF, Brott TG; CREST investigators. Influence of sex on outcomes of stenting versus endarterectomy: a subgroup analysis of the Carotid Revascularization Endarterectomy versus Stenting Trial (CREST). Lancet Neurol. 2011 Jun;10(6):530-7. doi: 10.1016/S1474-4422(11)70080-1. Epub 2011 May 5. PMID 21550314

RESULTS

PARTICIPANT FLOW:
Groups:
- Carotid-Artery Stenting (CAS): CAS involves insertion of a catheter or tube into an artery in the groin and then threading the catheter through the arteries of the body to the location of the plaque within the carotid artery in the neck. The stent is then placed to cover the plaque and hold the artery open.
Period: Overall Study
Arm/Group | Carotid-Artery Stenting (CAS) | Carotid Endarterectomy (CEA)
Started | 1262 | 1240
Completed | 1193 | 1129
Not Completed | 69 | 111
Not completed — Withdrawal by Subject | 36 | 64
Not completed — Lost to Follow-up | 33 | 47

BASELINE CHARACTERISTICS:
Groups:
- Carotid-Artery Stenting: Patients Randomized to CAS
- Carotid Endarterectomy: Patients Randomized to CEA
- Total: Total of all reporting groups
Arm/Group | Carotid-Artery Stenting | Carotid Endarterectomy | Total
Number analyzed (Participants) | 1262 | 1240 | 2502
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (9.0) | 69.2 (8.7) | 69.0 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 455 | 417 | 872
  Male | 807 | 823 | 1630
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 1172 | 1160 | 2332
  Non-White | 81 | 71 | 152
  Not Specified | 9 | 9 | 18
Symptomatic Status [Number; unit: Participants]
  Asymptomatic | 594 | 587 | 1181
  Symptomatic | 668 | 653 | 1321
Baseline Hypertension [Number; unit: Participants]
  Yes | 1080 | 1061 | 2141
  No | 179 | 172 | 351
  Unknown | 3 | 7 | 10
Diabetes Status [Number; unit: Participants]
  Yes | 384 | 375 | 759
  No | 873 | 857 | 1730
  Unknown | 5 | 8 | 13
Dyslipidemia [Number; unit: Participants]
  Yes | 1040 | 1053 | 2093
  No | 214 | 174 | 388
  Unknown | 8 | 13 | 21
Present Smoker [Number; unit: Participant]
  Yes | 329 | 317 | 646
  No | 915 | 899 | 1814
  Unknown | 18 | 24 | 42
Lesion Location [Number; unit: Participants]
  Left | 639 | 648 | 1287
  Right | 623 | 592 | 1215
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 141.6 (20.2) | 141.2 (20.5) | 141.4 (20.3)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 74.0 (11.6) | 73.9 (11.5) | 74.0 (11.5)
Percent Stenosis at Randomization [Number; unit: Participants]
  Moderate (<70%) | 165 | 186 | 351
  Severe (>=70%) | 1097 | 1054 | 2151

OUTCOME MEASURES:

1. Primary Outcome: Any Periprocedural Stroke, Myocardial Infarction, or Death During a 30-day Peri-procedural Period, and Postprocedural Ipsilateral Stroke Thereafter, up to 4-years.
Description: The primary aim of CREST is to assess if the efficacy of CAS differs from that of CEA in preventing stroke, myocardial infarction and death during a 30-day peri-procedural period, or ipsilateral stroke over the follow-up period in patients with symptomatic (>=50%) or asymptomatic (>=60%) extracranial carotid stenosis. Four-year follow-up, proportions reflecting the absolute efficacy of carotid-artery stenting (CAS) over that of carotid endarterectomy (CEA) were based on Kaplan-Meier survival estimates at the end of the 4 years.
Time Frame: 30 days and 4 years
Measure: Mean (Standard Error); unit: Percentage
Arm/Group | Carotid-Artery Stenting | Carotid Endarterectomy
Number analyzed (Participants) | 1262 | 1240
Percentage | 7.2 (0.8) | 6.8 (0.8)
Statistical Analysis 1: Comparison: Carotid-Artery Stenting vs Carotid Endarterectomy; Test type: Superiority or Other; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.81 to 1.51] — HR (95% CI) adjusted for age, sex and symptomatic status

2. Secondary Outcome: Differential Efficacy of CAS and CEA in Male and Female Participants in the Primary Endpoint (Any Periprocedural Stroke, Myocardial Infarction, or Death or Postprocedural Ipsilateral Stroke).
Description: 4-year follow-up, proportions reflecting the absolute efficacy of carotid-artery stenting (CAS) over that of carotid endarterectomy (CEA) were based on Kaplan-Meier survival estimates at the end of the 4 years.
Time Frame: 4 years
Measure: Mean (Standard Error); unit: Percentage
Arm/Group | Carotid-Artery Stenting | Carotid Endarterectomy
Number analyzed (Participants) | 1262 | 1240
Percentage
  Men | 6.2 (0.9) | 6.8 (1.0)
  Women | 8.9 (1.4) | 6.7 (1.3)
Statistical Analysis 1: Comparison: Carotid-Artery Stenting vs Carotid Endarterectomy; Test type: Superiority or Other; Hazard Ratio (HR) = 1.35, 95% CI 2-sided [0.82 to 2.23] — HR (95% CI) for WOMEN CAS vs CEA (adjusted for age and symptomatic status)

ADVERSE EVENTS:
Time Frame: Periprocedural period
Arm/Group | Carotid-Artery Stenting | Carotid Endarterectomy
Serious Adverse Events (participants affected / at risk) | 322/1262 | 292/1240
Other Adverse Events (participants affected / at risk) | 213/1262 | 212/1240
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carotid-Artery Stenting (N=1262) | Carotid Endarterectomy (N=1240)
Neurologic SAE (Nervous system disorders) | 98 (124) | 93 (108)
Hemorrhagic/Vascular SAE (Vascular disorders) | 32 (40) | 40 (53)
Hemodynamic SAE (Blood and lymphatic system disorders) | 73 (80) | 56 (63)
Infectious Disorder SAE (Infections and infestations) | 27 (31) | 19 (19)
Cardiovascular SAE (Cardiac disorders) | 36 (41) | 49 (58)
Angiographic/Procedural SAE (Surgical and medical procedures) | 9 (10) | 9 (11)
Miscellaneous SAE (General disorders) | 43 (50) | 47 (72)
Metabolic/Electrolyte SAE (Metabolism and nutrition disorders) | 4 (4) | 4 (4)
Other SAE (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carotid-Artery Stenting (N=1262) | Carotid Endarterectomy (N=1240)
Neurologic AE (non-endpoint, non-serious) (Nervous system disorders) | 65 (81) | 72 (83)
Hemorrhagic/vascular AE (not serious) (Vascular disorders) | 21 (23) | 20 (23)
Hemodynamic AE (not serious) (Blood and lymphatic system disorders) | 65 (73) | 45 (50)
Infectious Disorder AE (not serious) (Infections and infestations) | 13 (13) | 12 (13)
Cardiovascular AE (non-endpoint, non-serious) (Cardiac disorders) | 34 (41) | 36 (42)
Angiographic/Procedural AE (not serious) (Surgical and medical procedures) | 24 (27) | 43 (49)
Other AE (not serious) (General disorders) | 0 (0) | 1 (1)
Metabolic/Electrolyte AE (not serious) (Metabolism and nutrition disorders) | 8 (8) | 4 (4)
Miscellaneous Types of AEs (not serious) (General disorders) | 83 (132) | 86 (127)
Neurologic AE (endpoint, non-serious) (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No